CLINICAL TRIAL: NCT00280514
Title: Plasma and Abscess Fluid Pharmacokinetics of Cefpirome and Moxifloxacin After Single and Multiple Dose Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Markus Müller, Medical University of Vienna
Allocation: Non-Randomized
Other Study IDs: abscess-cef-moxi; EUdraCT no. 2005-004455-35
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2005-11

CONDITIONS: Abscess; Cysts
Keywords: abscess; penetration; antibiotics; cefpirome; moxifloxacin; abdominal cyst
MeSH Terms: conditions — Abscess; Cysts | interventions — Cefpirome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cefpirome and moxifloxacin administration

SUMMARY:
Penetration of cefpirome and moxifloaxacin into abscess fluid of humans will be tested. Patients with an abscess scheduled for drainage will receive study drugs (single or multiple dose), pus samples and plasma samples will be collected and analyzed by High pressure liquid chromatography (HPLC). Pharmacokinetics of the study drugs in pus and plasma will be determined using a pharmacokinetic model.

DETAILED DESCRIPTION:
Title: Plasma and abscess fluid pharmacokinetics of cefpirome and moxifloxacin single dose and multiple dose administration.

Background: Extensive research in the field of abscess treatment has established a claim for invasive drainage as the most efficient means of resolving suppurative lesions. In particular, computer tomography-guided percutaneous abscess drainage has repeatedly been reported to be advantageous compared to other invasive methods. However, application of the percutaneous interventional method is subject to some limitations. Coagulation abnormalities are considered a contraindication, and the absence of a safe anatomic access route, the presence of fistulas, severe inflammation of organs, or patients with advanced age have likewise been linked to low success rates of percutaneous abscess drainage. From these considerations, it becomes evident that percutaneous and surgical abscess drainage alone are not satisfactory in a number of patients suffering from abscess/infected cyst-related disease. In some patients antibiotic therapy is administered in bridging them to more stable conditions that drainage can be performed. Therefore, it is eminent for the overall outcome of patients to select an appropriate antibiotic. For this purpose, a model was recently developed to simulate the concentration time-curve of fosfomycin in abscess fluid after a single dose and after multiple doses.

Cefpirome and moxifloxacin are drugs which may be used in the empiric therapy of purulent infections. They may be used as monotherapy or they may be combined, e.g. with fosfomycin. Cefpirome is a 4th class cephalosporin with a broad spectrum (gram positive and gram negative pathogens), penetrating well into soft tissues. Moxifloxacin is a new fluoroquinolone with a considerable antimicrobial spectrum, also penetrating excellently into soft tissues. Based on the experiences with the methods and results obtained from our recent study on fosfomycin penetration into abscess fluid, the present pilot study will be set out to gain PK information on the penetration properties of cefpirome and moxifloxacin into abscess fluid and abdominal cysts.

Aim of the study: To determine pharmacokinetics of cefpirome and moxifloxacin in abscess (cyst) fluid and plasma after single and multiple doses.

Study design: Pharmacokinetic pilot study. Drug concentrations will be determined in abscess liquid upon drainage and in plasma over a period of eight hours.

Study population: 20 Patients with an abscess or an abdominal cyst, scheduled for surgical or computer tomography-guided drainage.

Methods: 1) High pressure liquid chromatography 2) Analysis of computer tomography (CT) images 3) Pharmacokinetic simulation model

Study drugs: Cefpirome (Cefrom, Aventis): will be administered to patients intravenously as single or multiple doses of 2 g dissolved in 100 mL of distilled water over 20 minutes. Moxifloxacin (Avelox, Bayer): will be administered to patients per os as tablet as single or multiple doses of 400 mg.

Patients: A total of 20 patients will be enrolled in the study. They will be assigned to 2 groups. Group 1: single dose (n = 12), Group 2: multiple doses (n = 8).

Main outcome variable: The cefpirome and moxifloxacin concentrations in abscess fluid will be measured. Considering plasma PK and the ratio of the surface to volume ratio of the abscess, the individual concentration-versus-time curve in abscess (cyst) fluid will be calculated. Individual pharmacokinetic parameters will be determined for abscess (cyst) fluid after a single dose and at steady state: AUC, AUC0-12/24h, Cmax, Tmax, t1/2ß, Cav(ss).

Additional outcome variables: Plasma (single dose and steady state): AUC, AUC0-12/24h, Cmax, Tmax, t1/2ß, Cav(ss). Pus and plasma: ratios of AUC and Cav(ss) to MIC, T>MIC The following parameters will be determined if possible: the diameter of the pericapsular space with enrichment of contrast agent, the degree of contrast agent enhancement in this zone and the pus density, rate of drug degradation in pus at body temperature in vitro, pH-value of pus, pus viscosity and specific weight.

Inconveniences and risks for patients:

The following side effects may occur after administration of cefpirome: Hypersensitivity reaction, allergic skin reactions, exanthema, urticaria, pruritus, drug fever, anaphylactic reactions, anaphylactic shock, interstitial nephritis, nausea, vomiting, abdominal pain, diarrhoea, pseudomembraneous colitis, elevation of liver enzymes and serum creatinine, thrombocytopenia, eosinophilia, hemolytic anemia, granulocytopenia, agranulocytosis, local irritation and pain at the site of injection, dysgeusia.

The following side effects may occur after administration of moxifloxacin:

Often or occasionally: Nausea, diarrhea, vomits, dyspepsia, QT-prolongation, elevation of AST, ALT, bilirubin, gamma GT, amylase, leucocytopenia, decrease of prothrombin, eosinophilia, thrombocythemia, thrombocytopenia, anemia, abdominal and head pain, dizziness, dysgeusia; unfrequent: asthenia, candidosis, thoracal and back pain, discomfort, leg pain, anaphylactic reactions, anaphylactic shock, insomnia, vortex, nervousness, tremor, paresthesia, discomposure, depression, hallucination, depersonalization, ataxia, xerostomia, flatulence, obstipation, anorexia, stomatitis, glossitis, tachycardia, edema, hypertension, palpitations, QT-prolongation, syncope, atrial fibrillation, angina pectoris, vasodilatation, hypotension, ventricular arrhythmia, torsade de pointe, hyperglycemia, hyperlipidemia, elevation of prothromin, icterus, arthralgia, myalgia, tendonitis, rash, pruritus, perspiration, urticaria, xerodermia, amblyopia, tinnitus, vaginitis, hepatitis, ataxia, tendon rupture, hypernatremia, hypercalcemia, neutropenia, hemolysis, transient loss of vision.

Total blood loss will be limited to a maximum of 85 mL, which is usually well tolerated by patients.

Risk/benefit assessment: CT and abscess drainage represent standard diagnosis and therapeutic procedures. Therefore, any risk associated with CT or abscess drainage is not ascribed to study procedures. Single and multiple doses of cefpirome (maximum of 14 doses) and moxifloxacin (maximum of 7 doses) are normally well tolerated and have very few side effects.

Ongoing therapy will not be affected or changed by study procedures. In summary, the risk conferred to patients by study procedures appears minimal.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, aged between 18 and 90 years.
* Written informed consent.
* Abscess formation or abdominal cyst scheduled to drainage.
* Plasma creatinine <1.5 mg/dL

Exclusion Criteria:

* Pregnancy or lactation.
* Hemodialysis or hemofiltration
* Allergy or hypersensitivity against study drugs
* Massive edemata or hypernatremia
* Reduced liver function (Child-Pugh A, B, C)
* Relevant prolongation of QT-interval
* CNS-diseases which predispose for cramps

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
AUC
AUC0-12/24h
Cmax
Tmax
t1/2ß
Cav(ss)

SECONDARY OUTCOMES:
ratios of AUC and Cav(ss) to MIC
T>MIC

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Pleiner, MD, Principal Investigator — Medical University of Vienna, Dep. of Clinical Pharmacology
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Sauermann R, Karch R, Langenberger H, Kettenbach J, Mayer-Helm B, Petsch M, Wagner C, Sautner T, Gattringer R, Karanikas G, Joukhadar C. Antibiotic abscess penetration: fosfomycin levels measured in pus and simulated concentration-time profiles. Antimicrob Agents Chemother. 2005 Nov;49(11):4448-54. doi: 10.1128/AAC.49.11.4448-4454.2005. PMID 16251282